CLINICAL TRIAL: NCT01124201
Title: Lumbar Segmental Stabilization, Strengthening and Stretching in Chronic Low Back Pain: a Comparative Study
Brief Title: Lumbar Stabilization, Strengthening and Stretching in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Fábio Jorge Renovato França, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1249/06
Record Dates: First submitted 2010-05-13; First posted 2010-05-14 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2007-03

CONDITIONS: Chronic Low Back Pain
Keywords: low back pain; clinical trial; stabilization; muscle stretching exercises; exercise therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Stabilization group (Experimental): In the Segmental Stabilization group exercises focused on the transversus abdominis and lumbar multifidus muscles.
  Interventions: Other: Stabilization , strengthening and stretching
- Strengthening group (Experimental): In the Superficial Strengthening group, exercises focused on the rectus abdominis, abdominus obliquus internus, abdominus obliquus externus and erector spinae muscles.
  Interventions: Other: Stabilization , strengthening and stretching
- Stretching group (Experimental): Stretching group: erector spinae, posterior connective tissues and ischiotibials muscles
  Interventions: Other: Stabilization , strengthening and stretching

INTERVENTIONS:
Other: Stabilization , strengthening and stretching — Interventions were conducted over 6 weeks, twice per week, lasting 30 minutes each. Sessions were supervised by the investigator, and participants were instructed to report any adverse event. Groups were instructed not to participate in any other physical program during the study. Forty-five patients were randomized into three groups namely: Segmental stabilization group (ES)(transversus abdominis and lumbar multifidus), superficial strengthening group (FS)(rectus abdominis, oblique abdominal muscles and erector spinae muscles) and stretching group (AL) (erector spinae, posterior connective tissues and ischiotibials muscles). Patients were evaluated for pain , functional disability,and ability to contract the TrA before and after the treatment.
  Other Names: Pressure Biofeedback Unit

SUMMARY:
The purpose of this study was to compare the efficacy of three exercise programs in patients with chronic low back pain: Segmental stabilization, superficial strengthening and stretching. Groups were contrasted regarding pain, functional disability and TrA muscle activation capacity. The three groups of exercise improved pain and functional disabilities, and the Segmental stabilization group was better in the ability to recruit TrA muscle.

DETAILED DESCRIPTION:
Objective: To contrast the efficacy of three exercise programs, segmental stabilization and strengthening of abdominal and trunk muscle and lumbar stretching on pain, functional impairment, and activation of the transversus abdominis muscle (TrA), in individuals with chronic low back pain.

Design: Forty-five patients were randomized into three groups namely: Segmental stabilization group (ES)(transversus abdominis and lumbar multifidus) (n=15, mean age 42,02 ± 8,15), superficial strengthening group (FS)(rectus abdominis, oblique abdominal muscles and erector spinae muscles) (n=15, mean age 41,71±6,41) and stretching group (AL) (erector spinae, posterior connective tissues and ischiotibials muscles) (n=15 mean age 41,53 ± 4,41). Groups were contrasted regarding pain (visual analogical scale and McGill pain questionnaire), functional disability (Oswestry disability questionnaire) and TrA muscle activation capacity (Pressure Biofeedback Unit = PBU). The program lasted 6 weeks, and sessions happened twice a week, with duration of 30 minutes each. Analysis of variance was used for inter and intragroup comparisons. Significance level was established at 5%.

Patients attended two weekly sessions during six weeks and were evaluated for pain (visual analogue scale and McGill Pain Questionnaire), functional disability (Oswestry disability index), and ability to contract the TrA (Pressure biofeedback unit) before and after the treatment. The treatment program consisted of 30 minutes sessions. The Anova one-way and Tukey´s Post Hoc were used to compare groups. The significance level adopted was 5%.

ELIGIBILITY:
Inclusion Criteria:

* low back pain for more than 3 months
* patients willing to participate and could participate in an exercise program safely and without cognitive impairments that would limit their participation.

Exclusion Criteria:

* past history of back surgery
* rheumatologic disorders
* spine infections
* spine exercise training in the 3 months before study onset.

Ages: 23 Years to 53 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2007-02; Primary Completion 2008-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Pain (visual analogical scale and McGill pain questionnaire) | Six weeks
Functional disability (Oswestry disability questionnaire) | Six weeks
TrA muscle activation capacity (Pressure Biofeedback Unit = PBU) | Six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fabio R França, MSc, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Barr KP, Griggs M, Cadby T. Lumbar stabilization: a review of core concepts and current literature, part 2. Am J Phys Med Rehabil. 2007 Jan;86(1):72-80. doi: 10.1097/01.phm.0000250566.44629.a0. PMID 17304690
- [Background] MacDonald DA, Moseley GL, Hodges PW. The lumbar multifidus: does the evidence support clinical beliefs? Man Ther. 2006 Nov;11(4):254-63. doi: 10.1016/j.math.2006.02.004. Epub 2006 May 23. PMID 16716640
- [Background] Ferreira PH, Ferreira ML, Maher CG, Refshauge K, Herbert RD, Hodges PW. Changes in recruitment of transversus abdominis correlate with disability in people with chronic low back pain. Br J Sports Med. 2010 Dec;44(16):1166-72. doi: 10.1136/bjsm.2009.061515. Epub 2009 May 26. PMID 19474006
- [Background] Liddle SD, Baxter GD, Gracey JH. Exercise and chronic low back pain: what works? Pain. 2004 Jan;107(1-2):176-90. doi: 10.1016/j.pain.2003.10.017. PMID 14715404
- [Background] Hayden JA, van Tulder MW, Malmivaara AV, Koes BW. Meta-analysis: exercise therapy for nonspecific low back pain. Ann Intern Med. 2005 May 3;142(9):765-75. doi: 10.7326/0003-4819-142-9-200505030-00013. PMID 15867409
- [Derived] Franca FR, Burke TN, Hanada ES, Marques AP. Segmental stabilization and muscular strengthening in chronic low back pain: a comparative study. Clinics (Sao Paulo). 2010;65(10):1013-7. doi: 10.1590/s1807-59322010001000015. PMID 21120303
- See also: Link to my thesis in portuguese. — http://www.teses.usp.br/teses/disponiveis/5/5163/tde-05032010-140030/